CLINICAL TRIAL: NCT05868785
Title: The Effect of Parenteral Nutrition During Nighttime Versus Daytime on Bone Turnover and Energy Metabolism in Intestinal Failure Patients
Brief Title: Effect of Nocturnal Parenteral Nutrition on Bone Turnover and Energy Metabolism
Acronym: NutriSync
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Mireille JM Serlie, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 82280.018.22
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Intestinal Failure; Osteoporosis; Insulin Sensitivity
Keywords: Parenteral Nutrition; Intestinal Failure; Circadian misalignment
MeSH Terms: conditions — Intestinal Failure; Osteoporosis; Insulin Resistance; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Intervention Model Description: Randomized crossover pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocturnal parenteral nutrition (Active Comparator): Patients will receive nocturnal parenteral nutrition, starting at 8pm
  Interventions: Dietary Supplement: Parenteral nutrition
- Diurnal parenteral nutrition (Experimental): Patients will receive diurnal parenteral nutrition, starting at 8am
  Interventions: Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Parenteral nutrition — Parenteral nutrition will be administered starting at 8 pm
  Other Names: active comparator
  Arms: Nocturnal parenteral nutrition
Dietary Supplement: Parenteral nutrition — Parenteral nutrition will be administered starting at 8 am
  Other Names: experimental
  Arms: Diurnal parenteral nutrition

SUMMARY:
This clinical trial will study the effect of daytime versus nighttime parenteral nutrition on bone turnover, glucose variability, nitrogen balance, sleep and wake rhythm and peripheral clock gene expression in patients with chronic intestinal failure.

DETAILED DESCRIPTION:
Objective: This randomized crossover pilot study aims to determine the effect of nocturnal versus daytime cyclic infusion of parenteral nutrition in adult patients with chronic intestinal failure on bone turnover, glucose metabolism, nitrogen balance, sleep and wake rhythm and clock genes expression.

This study will include 20 adult patients with chronic intestinal failure. Patients will receive nocturnal parenteral nutrition for 2 weeks (period A) and will switch to daytime parenteral nutrition (period B) for 2 weeks (random assignment). During both study periods glucose variability and sleep / wake rhythm will be measured. After both study periods, patients will be admitted to the metabolic unit for 24 hours to measure bone turnover markers, nitrogen balance, glucoregulatory hormones, energy expenditure and substrate oxidation rates and clock gene expression in leukocytes.

ELIGIBILITY:
Inclusion Criteria:

* Home parenteral nutrition for at least 5 nights a week
* On home parenteral nutrition for more than 1 year
* No major changes in parenteral nutrition for 3 months prior to inclusion

Exclusion Criteria:

* Parenteral infusion for more than 16 h a day
* Use of bone modifying drugs in the last 2 years
* Bone fractures in the past year
* Renal insufficiency (eGFR < 60 ml/min)
* HbA1c ≥48 mmol/ml
* Use of corticosteroids
* Shift work
* Performing intensive exercise (> 2 hours a day and > 3 times a week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Differences in bone turnover marker Procollagen 1 Intact N-Terminal Propeptide | Study day 1 versus study day 2
  Differences in the bone turnover marker Procollagen 1 Intact N-Terminal Propeptide (ug/L)
Differences in bone turnover marker carboxy-terminal collagen crosslinks | Study day 1 versus study day 2
  Differences in bone turnover marker carboxy-terminal collagen crosslinks (ng/L)
Changes in glucose variability | 2 weeks versus 2 weeks
  Changes in glucose variability measured by a continuous glucose monitor

SECONDARY OUTCOMES:
Changes in plasma insulin | Study day 1 versus study day 2
  insulin (pmol/L)
Changes in plasma glucagon | Study day 1 versus study day 2
  glucagon (ng/L)
Changes in nitrogen balance | Study day 1 versus study day 2
  Changes in nitrogen balance by comparing output (feces/urine) versus intake (oral/enteral/parenteral)
Changes in sleep/wake rhythm | 2 weeks versus 2 weeks
  Changes in sleep/wake rhythm measured by an actigraph
Changes in sleep quality | 2 weeks versus 2 weeks
  Changes in sleep quality, measured by Visual Analogue Scale (VAS) score (scale 1-10, higher scores mean better outcome)
Changes in clock gene expression | Study day 1 versus study day 2
  Changes in clock gene expression in leukocytes (if feasible; pilot)
Changes in energy expenditure | Study day 1 versus study day 2
  Changes in energy expenditure assessed by indirect calorimetry (kcal/24h)
Changes in substrate oxidation rates | Study day 1 versus study day 2
  Changes in substrate oxidation rates assessed by indirect calorimetry (percent)

OTHER OUTCOMES:
Changes in body temperature | Study day 1 versus study day 2
  Changes in body temperature measured by i-buttons (Celsius)

CONTACTS AND LOCATIONS:
Overall Officials: G.M. vd Werf, MSc, RD, Study Director — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be available after signing a data sharing agreement with the legal support office of the Amsterdam University Medical Center
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study results and for a period of 15 years
Access Criteria: Data sharing agreement with legal support office